CLINICAL TRIAL: NCT06708052
Title: Effects of Voodoo Flossing on Ankle Range of Motion, Balance, Gait Ability in Participants with Limited Ankle Dorsiflexion
Brief Title: Effects of Voodoo Flossing on Ankle in Participants with Limited Ankle Dorsiflexion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boung-hyoun Moon (Other Government)
Collaborators: Nambu University (Other Government)
Responsible Party: Sponsor-Investigator, Boung-hyoun Moon, Clinical Professor, Nambu University
Organization: Nambu University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1041478-2022-HR-008
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants Study
Keywords: voodoo flossing; limited ankle dorsiflexion
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Ankle application in voodoo flossing and control group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- voodoo flossing intervention (Experimental): The voodoo flossing intervention used the standard voodoo flossing, wrapping a voodoo flossing (lime green Sanctband Comprefloss™, 2" × 3.5 m; PENTEL, Shah Alam, Malaysia) made of natural rubber tightly around the ankle on the affected side. It was started at the fifth metatarsal and wrapped horizontally around the metatarsals twice, in a figure eight to the medial malleolus, over the Achilles tendon and the lateral malleolus three times, and around the medial malleolus again, before being passed twice from the medial mal-leolus over the Achilles tendon to the lateral malleolus, forming an end knot
  Interventions: Behavioral: voodoo flossing
- control (Sham Comparator): The control group did not use voodoo flossing.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: voodoo flossing — The voodoo flossing intervention used the standard voodoo flossing, wrapping a voodoo flossing (lime green Sanctband Comprefloss™, 2" × 3.5 m; PENTEL, Shah Alam, Malaysia) made of natural rubber tightly around the ankle on the affected side. It was started at the fifth metatarsal and wrapped horizontally around the metatarsals twice, in a figure eight to the medial malleolus, over the Achilles tendon and the lateral malleolus three times, and around the medial malleolus again, before being passed twice from the medial mal-leolus over the Achilles tendon to the lateral malleolus, forming an end knot
  Arms: voodoo flossing intervention
Behavioral: Control group — The control group did not use voodoo flossing.
  Arms: control

SUMMARY:
In the case of normal walking patterns, the angle of plantarflexion (PF) at heel contact should be 0 to 5 degrees, the angle of dorsiflexion (DF) in the terminal stance should be 10 degrees, and the angle of PF should be 15-20 degrees when the heel off. A therapist can apply a voodoo flossing to enhance range of motion (ROM), pain control, jumping performance, strength, myofascial release, and recovery from fatigue. This study compared the immediate effects of voodoo flossing application on ankle ROM, balance, and gait ability in stroke patients. Outcome measures were ankle ROM, weight bearing lunge test (WBLT) performance, static balance (one leg test), dynamic balance(Y-balance test) and gait ability. Outcome measures were assessed at baseline and immediately after applying the voodoo flossing.

DETAILED DESCRIPTION:
The voodoo flossing intervention used the standard voodoo flossing, wrapping a voodoo flossing (lime green Sanctband Comprefloss™, 2" × 3.5 m; PENTEL, Shah Alam, Malaysia) made of natural rubber tightly around the ankle on the affected side. It was started at the fifth metatarsal and wrapped horizontally around the metatarsals twice, in a figure eight to the medial malleolus, over the Achilles tendon and the lateral malleolus three times, and around the medial malleolus again, before being passed twice from the medial mal-leolus over the Achilles tendon to the lateral malleolus, forming an end knot. The participants were instructed to perform low-intensity active exercise involving ankle DF and plantar flexion for 2 minutes after applying the floss band. Then, the floss band was removed and the patient was asked to walk lightly on level ground for about 1 minute to allow reperfusion to normalize blood flow.

ELIGIBILITY:
Inclusion Criteria:

* less than 10° of dorsiflexion

Exclusion Criteria:

* lower extremity orthopedic problems
* unstable steps and balance
* visual impairments

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Ankle range of motion | 1 year
  Ankle passive ROM was measured using a universal goniometer in a non-weight bearing position. Subjects were prone with the knee joint at 90° . The ankle joint was set at 0° of eversion and inversion. The goniometer axis was placed beneath the lateral malleolus, and the stationary arm was positioned parallel to the fibula. The movable arm was positioned parallel to the fifth metatarsal, with the ankle in a neutral position. The measurement was repeated three times, and the average value was calculated. DF and PF measured angle.
Weight-bearing lunge test | 1 year
  The WBLT was performed to assess DF in a functional ankle joint. A measuring tape was placed horizontally on the floor perpendicular to a wall. The participants placed their affected-side foot on the tape with their big toe contacting the wall, and were instructed to touch the wall with the knee on the affected side. While maintaining this position, they were instructed to perform lunges by bending their knee, aiming for contact between their knee and the wall while keeping their heel firmly fixed on the floor. Once they were able to maintain knee and heel contact, the affected side foot was moved away from the wall, and they repeated the lunge test. The test was performed with 1-cm increases until knee and heel contact were no longer maintained. The maximum lunge distance was the far-thest distance from the wall to the big toe with the foot staying on the floor (without heel lifting) when the knee touched the wall. WBLT measured distance in centimeters.
Static balance ability | 1 year
  Static balance was assessed using the APDM Mobility Lab™ Opal inertial sensor system (APDM, Portland, OR, USA). The test was conducted in a quiet treatment room. During the test, participants were barefoot and wore three Opal inertial sensors: one over their clothing at the level of the fifth lumbar vertebra and one on each ankle. Each subject was instructed to maintain their balance as stably as possible in a barefoot one leg standing position for 30 seconds. The test was repeated three times at 30-second intervals. The static balance outcome measure was the postural sway area (cm/s2). The signal was sampled, processed automatically, and streamed to a laptop using Mobility Lab™ software (Mobility Lab, Arlington, VA, USA).
dynamic balance ability | 1 year
  The Y-Balance Test Lower Quarter (YBT-LQ; Move2Perform, Evansville, IN, USA) was used to assess dynamic ankle balance. The YBT-LQ device consists of three pipes extending from a central plate, each with a measurement indicator. The pipes are oriented in three directions: anterior (ANT), posterolateral (PL), and posteromedial (PM), forming angles of 135° between the anterior and posterior pipes and 90° between the posterior pipes. Each pipe is marked at 0.5 cm intervals. Participants stood on their measurement foot, aligning their big toe with the plate's red line, and reached maximally with the non-supporting foot to move the indicator along each pipe. The foot had to return to the starting position without losing balance or touching the ground. Incorrect attempts were repeated. The test recorded the indicator's distance, with each direction measured three times. Average values were calculated and normalized for analysis.
Gait ability | 1 year
  The APDM Mobility Lab™ Opal inertial sensor system (APDM) was used to assess gait based on the foot strike (FS) and toe-off (TO) angles. Data were collected from the sensor wirelessly at a sampling rate of 128 Hz and processed to quantify postural sway parameters. The test was conducted in a quiet treatment room. During the test, participants were barefoot and wore three Opal inertial sensors: one over their clothing at the level of the fifth lumbar vertebra and at each ankle. Verbal instructions were given to ensure accuracy. The subject was told to stand still at the start line until the first long tone was heard, at which time they started walking at a comfortable natural pace. When a second tone was heard after 2 minutes, the participants were asked to stop walking. After practicing for 30 seconds to become familiar with the test, participants were asked to walk back and forth along a straight 10-meter corridor at their usual pace for 2 minutes without a walking assist.

CONTACTS AND LOCATIONS:
Locations (1):
- Nambu University, Gwangju, Gwangsan-gu, South Korea

IPD SHARING:
Plan to Share IPD: No